# STATISTICAL ANALYSIS PLAN

A Phase 2, randomized, prospective, double-masked, vehicle-controlled study to assess the efficacy and safety of Nexagon® (NEXAGON) applied topically in subjects with corneal persistent epithelial defects (PED) resulting from severe ocular chemical and/or thermal injuries.

| Sponsor: | |
|-------------------|------------------|
| Protocol Number: | NEX-PED-005 |
| Author: | |
| Date:<br>Version: | 10FEB2022<br>1.0 |



| Protocol Number | er: NEX-PED-005 | |
|---|---|---|
| SAP Version: | 1.0 | |
| SAP Date: | 10FEB2022 | |
| Statistical Anal | ysis Plan Approval (Approval pg. 1 of 2 | 2) |
| | DocuSigned by: Rienne Leighton Signer Name: Rianna Leighton Signing Reason: I approve this document Signing Time: 10-Feb-2022 15:25 CST CD94786303324D1CB8620BDCA6E60A71 | |
| Prepared by:<br> <br> <br> <br> | | 10-Feb-2022 15:25 CST Date |
| | DocuSigned by: Garrick Wallstrom Signer Name: Garrick Wallstrom Signing Reason: I approve this document Signing Time: 10-Feb-2022 18:19 EST DE0A4A68DA3E4AC08AD3A5675C82F53D | 10-Feb-2022 18:19 EST |
| Reviewed by:<br> <br> <br> <br> | | Date |

# Statistical Analysis Plan Approval (Approval pg. 2 of 2)



#### **Table of Contents**

| Table | of Contents | 4 |
|---|---|---|
| List of | Abbreviations | 7 |
| 1. | Introduction | S |
| 2. | Study Objectives | 9 |
| 2.1 | Primary Endpoint | 9 |
| 2.2 | Secondary Endpoints | 9 |
| 2.3 | Exploratory Endpoints | 9 |
| 2.4 | Safety Variables | 10 |
| 2.5 | Statistical Hypotheses | 10 |
| 3. | Study Design and Procedures | 11 |
| 3.1 | General Study Design | 11 |
| 3.2 | Study Visit Windowing | 13 |
| 3.3 | Dose Regimen, Study Flow Diagram, and Schedule of Visits and Assessments | 17 |
| 4. | Study Treatments | 23 |
| 4.1 | Method of Assigning Subjects to Treatment Groups | 23 |
| 4.2 | Masking and Unmasking | 23 |
| 5. | Sample Size and Power Considerations | 23 |
| 6. | Data Preparation | 24 |
| 6.1 | Input Data | 24 |
| 6.2 | Output Data | 24 |
| 7. | Analysis Populations | 25 |
| 8. | General Statistical Considerations | 26 |
| 8.1 | Unit of Analysis | 26 |
| 8.2 | Missing or Inconclusive Data Handling | 26 |
| 8.3 | Definition of Baseline and Final On-Treatment Visit | 27 |
| 8.4 | Data Analysis Conventions | 28 |
| 8.5 | Adjustments for Multiplicity | 28 |
| 9. | Disposition of Subjects | 29 |
| 10. | Demographic and Pretreatment Variables | 30 |
| 10. | 1 Demographic Variables | 30 |

| 10.2 | 2 Pretreatment Variables | 30 |
|---|---|---|
| 11. | Medical History and Concomitant Medications | 31 |
| 11.1 | 1 Medical History | 31 |
| 11.2 | 2 PED History | 31 |
| 11.3 | 3 Prior and Concomitant Medications | 31 |
| 11.4 | 4 Concomitant Procedures | 32 |
| 12. | Treatment Exposure | 32 |
| 13. | Efficacy Analyses – Masked Portion of Study | 32 |
| 13.1 | 1 Primary Efficacy Outcome Analysis | 32 |
| 1: | 3.1.1 Sensitivity Analyses | 34 |
| 13.2 | 2 Secondary Efficacy Outcome Analyses | 34 |
| 13 | 3.2.1 Time to Corneal Epithelial Recovery | 35 |
| 13 | 3.2.2 Visual Acuity | 35 |
| 13 | 3.2.3 Number of Treatment Doses | 36 |
| 14. | Exploratory Analyses | 36 |
| 14.1 | 1 Change from Baseline in PED Area | 37 |
| 14.2 | 2 Corneal Re-epithelialization | 37 |
| 14.3 | 3 Change from Baseline in Ocular Symptoms | 37 |
| 14.4 | 4 Open-Label Analyses for Subjects Receiving Salvage Dose | 39 |
| 14.5 | 5 Intra-Subject Corneal Re-epithelialization in Fellow Eye of Subjects with Bilateral Inju | ıries40 |
| 15. | Safety Analyses | 40 |
| 15.1 | 1 Adverse Events | 40 |
| 15.3 | 3 Slit Lamp Examination | 43 |
| | 4 PED Assessment Including Digital Photography | |
| | 5 Ophthalmoscopy | |
| 15.6 | 6 Intraocular Pressure | 45 |
| 15.7 | 7 Clinical Laboratory Data | |
| 16. | Interim Analyses | 46 |
| 16.1 | 1 IA Stage 1 | 46 |
| 16.2 | 2 IA Stage 2 | 48 |
| 17. | Changes from Protocol-Stated Analyses | 50 |
| 18. | References | 50 |
| 19. | Revision History | 50 |
| | Revision Flistory | |

| 21. | Tables for Interim Analyses | 54 |
|-----|-----------------------------|----|
| 22. | Data Listings | 57 |
| 23 | Figures | 59 |



| ADaM | Analysis Data Model |
|----------|----------------------------------------------|
| AE | Adverse Event |
| ANCOVA | Analysis of Covariance |
| ATC | Anatomical Therapeutic Chemical |
| BCVA | Best Corrected Visual Acuity |
| CF | Counting Fingers |
| CI | Confidence Interval |
| COVID-19 | Coronavirus (COVID-19) pandemic |
| CP | Conditional Power |
| CRA | Clinical Research Associate |
| CRO | Contract Research Organization |
| CS | Clinically Significant |
| DTA | Data Transfer Agreement |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| EOS | End of Study |
| ETDRS | Early Treatment Diabetic Retinopathy Study |
| FAS | Full Analysis Set |
| FAS-IA | Full Analysis Set for the IA |
| FUP | Follow-up |
| HM | Hand Movements |
| IAP1 | Interim Analysis Primary Endpoint 1 |
| IAP2 | Interim Analysis Primary Endpoint 2 |
| IAS1 | Interim Analysis Secondary Endpoint 1 |
| IAS2 | Interim Analysis Secondary Endpoint 2 |
| ICH | International Conference on Harmonisation |
| IOP | Intraocular Pressure |
| LOCF | Last Observation Carried Forward |
| logMAR | Logarithm of the Minimum Angle of Resolution |
| LS | Lease Squares |
| IP | Investigational Product |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NCS | Not Clinically Significant |
| NPL | No Perception of Light |
| OL | Open-Label |
| PCI | Potentially Clinically Important |
| PDF | Portable Document Format |
| PED | Persistent Epithelial Defect |
| PL | Perception of Light |
| PP | Per Protocol |
| PT | Preferred Term |
| re-epi | re-epithelialization |

| RTF | Rich Text Format |
|---------|-------------------------------------------|
| SaaS | Software-as-a-Service |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDC | Statistics & Data Corporation |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| TEAE | Treatment-Emergent Adverse Event |
| VA | Visual Acuity |
| WHODrug | World Health Organization Drug Dictionary |

#### 1. Introduction

The purpose of this statistical analysis plan (SAP) is to describe the planned analyses and reporting for protocol NEX-PED-005,

This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials and the most recent ICH E3 Guideline, entitled Guidance for Industry: Structure and Content of Clinical Study Reports.

This SAP describes the data that will be analyzed and the subject characteristics, efficacy, and safety assessments that will be evaluated. This SAP provides details of the specific statistical methods that will be used. The statistical analysis methods presented in this document will supersede the statistical analysis methods described in the clinical protocol, and any changes to the protocol stated analyses will be detailed in Section 17. If additional analyses are required to supplement the planned analyses described in this SAP, they may be completed and will be identified in the clinical study report.

#### 2. Study Objectives

The objective of this study is to assess the efficacy and safety of two topical ocular dose concentrations of Nexagon® (NEXAGON) as a treatment for non-healing corneal persistent epithelial defects (PEDs) resulting from severe chemical and/or thermal ocular injuries.

#### 2.1 Primary Endpoint

The primary efficacy endpoint is corneal epithelial recovery, defined as a cornea that re-epithelializes by of treatment and remains re-epithelialized for after initial re-epithelialization was first recorded, as assessed by the Investigator.

#### 2.2 Secondary Endpoints

#### 2.3 Exploratory Endpoints



#### 2.4 Safety Variables

The safety variables include the incidence of treatment-emergent adverse events (TEAEs).

#### 2.5 Statistical Hypotheses

The null and alternative hypotheses, based on the primary endpoint, are as follows:





#### 3. Study Design and Procedures

#### 3.1 General Study Design

This phase 2 multi-center trial is a randomized, prospective, double-masked, vehicle-controlled study to assess the efficacy and safety of NEXAGON applied topically in subjects with corneal PED resulting from severe ocular chemical and/or thermal injuries.

A subject's participation is to start with screening (Eligibility Assessment Visit) to determine eligibility for enrollment into the study prior to Day 1. If the subject is considered eligible for the study, the subject will be randomized to receive either NEXAGON or NEXAGON or Vehicle , respectively on Day 1.

For all subjects, the first investigational product application will occur following randomization with investigational product (NEXAGON or NEXAGON

| | or Vehicle) |
|---|---|
| | . Following investigational product application, |
| | tudy will comprise of 2 periods,a Treatment Period and Post-healing Follow-up Period: reatment Period (Masked): |
| | uring the Treatment Period, masked investigational product will be administered on |
| - | If re-epithelialization of the defect has NOT occurred another single application of masked investigational product will be administered |
| - | If re-epithelialization occurs at any time during the masked Treatment Period, subjects will enter a Post-healing Follow-up Period to assess durability of the corneal epithelium. |
| - | |
| P | ost-healing Follow-up Period (Masked) |
| | uring the Post-healing Follow-up Period subjects will be assessed lower |
| - | If the healed epithelium is sustained within the Post-healing Follow Period (durable), the subject will then exit the study having completed all visits. |
| - | |
| 0 | pen-Label Section |
| In | the open-label section of the study subjects will receive a salvage dose of NEXAGON |
| - | If re-epithelialization has not been achieved dose of |
| | NEXAGON will be applied A final assessment of healing for these subjects will be conducted |
| - | |

#### 3.2 Study Visit Windowing

Study day will be referred to in all tables and listings. Table 1a shows the planned study visits and the acceptable visit window for each visit for subjects who are in the study for the maximum duration. Table 1b shows the planned study visits and acceptable visit window by study period. Visits that are not able to be completed within the windows specified in the protocol must be recorded as protocol deviations.

Note: Day 1 corresponds to the day of randomization, there is no Day 0.

following the final application of investigational product.





Table 1b. Study Visit Windows





The dosing regimen is provided in Figure 1, the study flow diagram (visit schedule and dosing days) is provided in Figure 2 and the schedule of visits and assessments is provided in Table 2.



Figure 2. Study Flow Diagram –



#### 4. Study Treatments

#### 4.1 **Method of Assigning Subjects to Treatment Groups**

A subject who meets all the inclusion criteria and none of the exclusion criteria is eligible for randomization Subjects are to be randomized to one of three treatment group:

| | <ul> <li>GROUP A – NEXAGON</li> <li>GROUP B – NEXAGON</li> </ul> |
|---|---|
| | • GROUP C – Vehicle (0%) |
| | A statistician not directly involved in the analysis of the study results will prepare the randomization schedule using block randomization to maintain balance between treatment groups. Randomization is to be done |
| | When a subject is confirmed to be eligible for randomization treatment assignment for that subject will be determined by |
| 4.2 | Masking and Unmasking |
| | All subjects, investigators, and study personnel involved with the conduct of the study will be masked with regard to treatment assignments. |
| | The Investigator may unmask a subject's treatment assignment only in the case of an emergency when knowledge of the investigational product is essential for the clinical management or welfare |
| | of the subject. |
| | If a drug-related serious adverse event (SAE) is reported, the Medical Monitor may unmask the treatment assignment for the individual subject. |
| 5. | Sample Size and Power Considerations |
| | Assuming the true rate of corneal epithelialization in each of the NEXAGON arms of |
| | Assuming a discontinuation rate |
| | Enrollment will continue until |

#### 6. Data Preparation

#### 6.1



6.2



| | Define.xml will be created for SDTM and ADaM |
|----------|----------------------------------------------|
| 7. Analy | rsis Populations |
| _ | |

| 8. | Gen | eral Statistical Considerations |
|-----|-----|---------------------------------------|
| 8.1 | | Unit of Analysis |
| | | The study eye will be defined as |
| 8.2 | | Missing or Inconclusive Data Handling |

| Protoc | ol NEX-PED-005 SAP, Version 1.0 |
|---|---|
| 8.3 | Definition of Baseline and Final On-Treatment Visit Baseline will be defined as the last measurement prior to the first dose of study medication. Change from baseline will be calculated as follow-up visit value minus baseline value. |
| | enange nem zassime wii ze salealatea as tellen ap violi value minus zassime value. |
| | The final on-treatment visit is defined as the day of initial corneal re-epithelialization, treatment or day of discontinuation during treatment. |

# 8.4 Data Analysis Conventions

All data analysis will be performed by after the study is completed and the database has been locked and released for unmasking. Statistical programming and analyses will be performed using Output will be provided in rich text format (RTF) for tables and portable document format (PDF) for tables, listings, and figures using landscape orientation. All study data will be listed by subject, treatment, and visit (as applicable) based on all randomized subjects unless otherwise specified.

Summaries for continuous and ordinal variables will include the number of observations (n), arithmetic mean, standard deviation (SD), median, minimum, and maximum. Minima and maxima will be reported with the same precision as the raw values; means and medians will be presented to one additional decimal place than reported in the raw values. Standard deviations will be presented to two additional decimal places than reported in the raw values. Summaries for discrete variables will include counts and percentages. All percentages will be rounded to one decimal place (i.e., XX.X%). Differences between active treatment groups and placebo will be calculated as active minus placebo and change from baseline will be calculated as follow-up visit minus baseline.

| • | • | • |
|---|---|---|

Unless otherwise specified, summaries will be presented by treatment group and, where appropriate, visit. Listings will be sorted by treatment group, subject number, visit/time point, and parameter as applicable.

# 8.5 Adjustments for Multiplicity



| Pro | otocol NEX-PED-005 SAP, Version 1.0 |
|---|---|
| 9. | Disposition of Subjects Subject enrollment, inclusion in analysis populations, and study completion/withdrawal from the study for the main study as well as the open-label section of the study will be summarized and listed in terms of the numbers and percentages of subjects who were randomized, completed the study, and discontinued from the study. Subjects who are not discontinued from the study will be considered study completers. Disposition will be summarized by treatment group and for all subjects. |
| | The number and percentage of subjects prematurely discontinued from the study and the reasons for study discontinuation will be summarized by treatment group for all subjects who discontinued the study. The reasons for study discontinuation that will be summarized include AE, lost to follow-up physician decision, protocol violation, screen failure, study terminated by sponsor, withdrawal by subject, and other. |
| | The number and percentage of subjects with major protocol deviations will be summarized by treatmen group for all randomized subjects. |

| de age, gender at birth, race, and ethnicity |
|----------------------------------------------|
| s will be provided. |
| eparately for all randomized subjects |

Summaries will be presented for the study eye. For subjects with a bilateral ocular injury, the assessments detailed above will also be listed for the fellow eye (in addition to the study eye).

# 11. Medical History and Concomitant Medications

### 11.1

11.2

11.3

| Medical History |
|---|
| General ocular history, and non-ocular medical history will be coded using the Medical Dictionary |
| for Regulatory Activities (MedDRA) Medical history, including details of any ongoing |
| medical conditions, will be recorded prior to Day 1 and before eligibility is confirmed. |
| SOCs will be listed in alphabetical order and PTs within an SOC will be listed in order of descending frequency across all subjects. |
| Listings of medical history will be generated separately for both ocular data and non-ocular data. |
| PED History |
| A detailed ocular examination and history will be conducted prior to the Day 1 visit and assessed |
| against the inclusion and exclusion criteria of the protocol. |
| Prior and Concomitant Medications |

| Protoc | col NEX-PED-005 SAP, Version 1.0 |
|---|---|
| | Prior and concomitant medications will be listed for all randomized subjects. |
| | The and concernate medications will be listed for all randomized casjects. |
| 11.4 | Concomitant Procedures |
| | Concomitant procedures will be coded using the Medical Dictionary for Regulatory Activities |
| | (MedDRA) and summarized by SOC and PT. |
| | Concomitant procedures will be listed using all randomized |
| | Concomitant procedures will be listed using all randomized |
| 12. T | reatment Exposure |
| | Treatment exposure will be defined in two ways, as the extent of treatment exposure and the |
| | number of treatment doses. The number of treatment doses is the number of actual applications |
| | of NEXAGON or Vehicle. |
| | fficacy Analyses – Masked Portion of Study |
| 13.1 | Primary Efficacy Outcome Analysis |
| | The primary efficacy outcome will be the comparison of each dose of NEXAGON to Vehicle for |
| | the proportion of subjects with corneal epithelial recovery, defined as a cornea that re-epithelializes |
| | of treatment and remains re-epithelialized after initial re-epithelialization |
| | was first recorded (during the masked treatment portion of the study and assessed by the |



The number and proportion of subjects with corneal epithelial recovery will be summarized by treatment group and tested between treatment groups

# Protocol NEX-PED-005 SAP, Version 1.0 The following secondary efficacy endpoints, 13.2.1

| Exploratory Analyses The exploratory efficacy outcomes will be | | | | |
|---|---|---|---|---|
| Exploratory Analyses The exploratory efficacy outcomes will be | | | | |
| Exploratory Analyses The exploratory efficacy outcomes will be | _ | | | |
| Exploratory Analyses The exploratory efficacy outcomes will be | _ | | | |
| Exploratory Analyses The exploratory efficacy outcomes will be | | | | |
| The exploratory efficacy outcomes will be | | | | |
| The exploratory efficacy outcomes will be | -<br>- | v Analyses | | |
| | | | cv outcomes wil | l he |
| | THE 67 | Apioratory officat | sy catoomice wii | |
| | _ | | | |


an already present event that worsens either in intensity or frequency following treatment.

be recorded from the time of first application of the investigational product and until the final visit.

Treatment-emergent adverse events (TEAEs), defined as AEs that occur after the first dose of study medication, are undesirable events not present prior to investigational product treatment, or

Serious Adverse Events (SAE) any untoward medical occurrence that at any dose results in death, is life-threatening and/or sight threatening, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect. SAEs are undesirable events (experiences) or reaction not present prior to investigational product treatment, or an already present event that worsens in magnitude to be classified as an SAE, either in intensity or frequency following treatment.

Severity of an AE is defined as a qualitative assessment of the degree of intensity of an AE as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of relationship to study drug or seriousness of the event and should be evaluated according to the following scale:

- Mild: Event is noticeable to the subject but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate: Event is bothersome, possibly requiring additional therapy, and may interfere
  with the subject's daily activities.
- Severe: Event is intolerable, necessitates additional therapy or alteration of therapy, and interferes with the subject's daily activities.

The relationship of each AE or SAE to the study drug should be determined by the Investigator using these explanations: definitely related, probably related, possibly related, unlikely to be related, and unrelated. Only definitely, probably, and possibly related TEAEs will be considered as treatment-related TEAEs. For TEAEs prior to rescue medication use, only those TEAEs with an onset date prior to the date that rescue medications were first used will be included.

Clinically significant abnormal laboratory findings or other abnormal assessments that are present at baseline and significantly worsen following the start of the study will be reported as AEs and SAEs. The Investigator will exercise his/her medical and scientific judgment in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant.

Verbatim descriptions of AEs will be mapped to MedDRA terms and presented in a data listing. Adverse events recorded in the eCRF which began prior to treatment will not be included in the summary tables but will be included in the AE data listings. All AEs, SAEs, and TEAEs will be presented separately in subject data listings. The TEAEs leading to study treatment discontinuation will also be listed separately.

An overall summary will be presented that includes the number of events and the number and percentage of subjects who experienced at least one TEAE, by treatment group and over all subjects. This summary will also include breakdowns of TEAEs further categorized as ocular (study eye and, for subjects with bilateral injury, fellow eye separately) or non-ocular, treatment-related TEAEs, TE-SAEs, TEAEs leading to treatment withdrawal, TEAEs leading to death, TEAEs by maximal severity, and TEAEs by relationship to study drug.

Treatment-emergent adverse events (TEAEs), those that occur after the first dose of study medication, will be summarized by treatment group using frequency and percentages for each SOC and PT within each SOC. Similar summaries will be presented for treatment related TEAEs, TEAEs by maximum severity, serious TEAEs, and TEAEs leading to test article discontinuation.

Separate summaries of TEAEs will be provided showing the number and percentage of subjects who experienced at least one TEAE by treatment group and over all subjects. Non-ocular TEAEs will be summarized using discrete summary statistics and presented by treatment group at the subject and event level by SOC and PT. Ocular TEAEs will be similarly summarized at the subject level for study and fellow eyes separately. If a subject reports the same PT multiple times within the same SOC, that PT will only be reported once within that SOC. As with the PT, if a subject reports multiple conditions within the same SOC, that SOC will only be reported once. In the summary, SOCs will be listed in ascending alphabetical order; PTs will be listed in order of descending frequency for all subjects within each SOC.

The number of subjects with any TEAEs (along with percentages) will be tabulated by SOC and PT within each SOC by treatment group. Summaries of TEAEs by maximal severity, strongest relationship to study drug, and strongest relationship to study drug and maximal severity will be presented for ocular AEs and non-ocular AEs separately. To count the number of subjects with any TEAEs, if a subject has multiple TEAEs coded to the same PT within the same SOC, the subject will be counted once under the maximum severity. TEAEs that led to test article discontinuation, defied as drug interruption or drug withdrawal as response to the AE, treatment related TEAEs, and TE-SAEs will also be summarized by SOC and PT.

| Protoco | EX-PED-005 SAP, Version 1.0 | |
|---|---|---|
| 15.4 | ED Assessment | |
| 10.4 | e epithelial defect size will be assessed prior to Day 1 and randomization on Day 1 the | n at each |
| | low-up visit. | |
| 15.5 | | |

No specific laboratory results (other than a positive pregnancy test) will be used to exclude a subject from entry or continued participation in the study, unless in the Investigator's opinion the results indicate the subject has a concurrent condition that may affect the safety of the subject or potentially the outcome of the study.

| The same blood tests will be repeated when the subject completes the Treatment Period of th |
|---|
| study. Refer to Table 2 (Schedule of Assessments). |

Laboratory data will be presented in data listings. Clinical laboratory results will be summarized using continuous summaries, including continuous change from baseline. Qualitative laboratory values will be summarized with discrete statistics, including frequency and percent of subjects with normal, abnormal, high, and low values and using shift tables from baseline. A listing of potentially clinically important (PCI) laboratory findings will also be presented, where PCI is defined as any laboratory results that are abnormal, high or low.

| 16. |
|-----|

| Protoco | I NEX- | PED-005 SA | P, Version 1 | 1.0 | | | |
|---------|--------|------------|--------------|-----|---|---|------|
| | _ | | | | | | |
| | i | | | | I | | |
| ļ | | | | | | | |
| ļ | | | | | | | |
| 16.2 | | | | | | | |
| 10.2 | | | | | | | |
| | | | | | | _ | |
| | _ | | | | | | |
| | • | | | | | | |
| | | | | | | 1 | |
| | | | | | | | <br> |
| | | | | | | | <br> |





#### 18. References

- 1. Brookmeyer R, Crowley J. A confidence interval for the median survival time. *Biometrics*. 1982;38:29-41.
- 2. Chan, I. S. F., and Zhang, Z. (1999). "Test-Based Exact Confidence Intervals for the Difference of Two Binomial Proportions." Biometrics 55:1202–1209.

### 19. Revision History

Documentation of revision to the SAP will commence after approval of the final version 1.0.

#### 20. Tables for Final Analysis

Tables that will be included in the topline delivery are shown in boldface font.

| T 11 N | | 2 14 |
|--------------|-----------------------------|-------------------------|
| Table Number | Title | Population |
| 14.1.1 | Subject Disposition | All Randomized Subjects |
| 14.1.2.1.1 | Demographic Characteristics | All Randomized Subjects |
| 14.1.3.1 | Ocular Medical History | Safety Population |
| 14.2.1.1 | Corneal Epithelial Recovery | Full Analysis Set |



| | Overall Summary of TEAEs by Treatment | |
|----------|------------------------------------------|-------------------|
| 14.3.1 | Group | Safety Population |
| | Ocular TEAEs by System Organ Class and | |
| 14.3.2.1 | Preferred Term (Study Eye) | Safety Population |
| | TEAEs That Led to Premature Test Article | |
| 14.3.6 | Discontinuation | Safety Population |



### 21. Tables for Interim Analyses

Tables that will be included in Interim Analysis Stage I are shown in boldface font.

| Table Number | Title | Population |
|--------------|-------|------------|
| 1 | | |
| • | | |
| _ | | |
| · | | |





# 22. Data Listings

| Listing<br>Number | Title | Population |
|-------------------|------------------------|-------------------------|
| 16.1.7 | Randomization Schedule | All Randomized Subjects |
| 16.2.1.1 | Subject Disposition | All Randomized Subjects |

| 16.2.2.1 | Protocol Deviations | All Randomized Subjects |
|---|---|---|
| 16.2.4.1 | Demographics | All Randomized Subjects |
| 16.2.4.2.1 | Ocular Medical History | All Randomized Subjects |
| 16.2.4.2.2 | Non-Ocular Medical History | All Randomized Subjects |
| 16.2.4.3 | PED History | All Randomized Subjects |
| 16.2.4.4 | Ocular Prior and Concomitant Medications | All Randomized Subjects |
| | Non-Ocular Prior and Concomitant | |
| 16.2.4.5 | Medications | All Randomized Subjects |
| 16.2.4.6 | Concomitant Procedures | All Randomized Subjects |
| 16.2.5 | Investigational Product Administration | All Randomized Subjects |
| 16.2.7.1 | All Adverse Events | All Screened Subjects |
| 16.2.7.2.1 | Treatment-Emergent Adverse Events | All Screened Subjects |
| | Treatment-Emergent Adverse Events | |
| 16.2.7.2.2 | Leading to Test Article Discontinuation | All Screened Subjects |
| | Treatment-Related Treatment-Emergent | |
| 16.2.7.2.3 | Adverse Events | All Screened Subjects |
| 16.2.7.3 | Serious Adverse Events | All Screened Subjects |
| 40.0.5 | Clinical Laboratory Measurements – | |
| 16.2.8.1.1 | Hematology | All Randomized Subjects |



## 23. Figures

| Figure<br>Number | Title | Population |
|------------------|-------|------------|